CLINICAL TRIAL: NCT07074496
Title: An Open, Prospective, Single-arm Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of Allogeneic Anti CD19 CAR-T Combined With a Novel Third-generation TKI Olverembatinib in Patients With Newly Diagnosed Philadelphia Chromosome-Positive Acute Lymphoblastic Leukemia.
Brief Title: Efficacy, Safety, and Pharmacokinetics of ThisCART19A Combined With Olverembatinib in Patients With Newly Diagnosed Philadelphia Chromosome-Positive Acute Lymphoblastic Leukemia.
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: Fundamenta Therapeutics, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ThisCART19A Ph+ALL
Record Dates: First submitted 2024-01-06; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Philadelphia Chromosome-Positive Acute Lymphoblastic Leukemia
MeSH Terms: interventions — fludarabine; Cyclophosphamide; olverembatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Group (Experimental): ThisCART19A cells infusion, Given intravenously，Combined With Olverembatinib, Given PO
  Interventions: Drug: ThisCART19A; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Olverembatinib

INTERVENTIONS:
Drug: ThisCART19A — ThisCART19A is a new type CAR-T therapy for patients with ph+ ALL.
Drug: Fludarabine — Fludarabine is used for lymphodepletion.
Drug: Cyclophosphamide — Cyclophosphamide is used for lymphodepletion.
Drug: Olverembatinib — a third-generation TKI

SUMMARY:
This is an Open, Prospective, Single-arm Study, which is designed to evaluate the efficacy, safety and pharmacokinetics of ThisCART19A Combined With Olverembatinib for the treatment of Newly Diagnosed Ph-positive lymphoblastic leukemia.

DETAILED DESCRIPTION:
To evaluate the efficacy, safety and pharmacokinetics of ThisCART19A Combined With Olverembatinib for the treatment of Ph-positive lymphoblastic leukemia. Newly diagnosed Ph-positive patients will be given VP chemotherapy for induction treatment until the leukocyte count is less than 10×109/L. Then chemotherapy regimen of fludarabine and cyclophosphamide followed by a infusion of ThisCART19A. These patients will combination with Olverembatinib as maintenance therapy based on the hematologic complete remission of leukemia after 4 weeks of treatment.

Patients could receive an additional infusion of ThisCART19A if they achieved initial benefit and subsequently minimal residual disease positive (defined as Flow-cytometric MRD≥0.1%) during maintenance treatment. Additionally, a subset of patients which achieved complete molecular remission over 6 month were eligible for a second planned infusion as a consolidation therapy .

During the treatment, lumbar puncture combined with sheath injection will be performed to prevent central nervous system leukemia (CSNL). If CNSL occurs at the time of admission, patients should receive regular conventional lumbar puncture and sheath injection for treating CNSL.

During the treatment, each subject will be evaluated regularly, including hematological response, FCM-MRD, cytogenetic response and molecular remission rate, as well as adverse events. EFS and OS will be followed up for 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non-lactating female patients who are 18 years of age or older.
2. Newly diagnosed Philadelphia chromosome-positive (Ph+) or BCR-ABL1-positive ALL, as defined by the 2016-WHO criteria. Participants should not be treated with any kind of TKIs or chemotherapy.
3. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2, and expected survival period ≥ 3 months.
4. Organ function as indicated by the following laboratory indicators must be met:

1. Alanine aminotransferase (ALT) ≤ 5×upper limit of normal (ULN), aspartate aminotransferase (AST) ≤ 5×ULN; 2. Total bilirubin<2×ULN; 3. 24-hour calculated creatinine clearance>30 mL/min; 4. SpO2≥92%; 5. Cardiac ejection fraction (EF)≥40%;

Exclusion Criteria:

1. Active hepatitis B virus (defined as serum HBV-DNA ≥ 2000 IU/mL), hepatitis C virus (HCV), human immunodeficiency virus (HIV) or active syphilis infection prior to enrollment. (Subjects with HBV-DNA < 2000 IU/mL can be enrolled, but should be administered antiviral drugs such as entecavir and tenofovir with relative clinical indicators monitored simultaneously during the treatment.) ;
2. Uncontrolled active infection;
3. Patients who are currently suffering from active autoimmune disease or a history of autoimmune disease potentially involving the CNS;
4. Patients who have any history of heart or vascular disease, such as hypertension (systolic blood pressure(HBP) > 140mmHg and/or diastolic blood pressure > 90mmHg);
5. Cardiac ultrasonography indicates that pulmonary artery systolic blood pressure is >50 mmHg; or there are clinical symptoms related to pulmonary arterial hypertension;
6. Patients who suffer from severe bleeding disorders unrelated to Ph+ ALL;
7. Patients who have any other malignant tumors that require treatment;
8. Patients who have severe hypertriglyceridemia (triglyceride ≥ 5.6mmol/L);
9. Patients who are pregnant, planning to become pregnant or breastfeeding;
10. Patients who underwent major surgery (except for minor surgery such as catheter placement or bone marrow biopsy) within 14 days before the first drug;
11. Patients who may not be able to complete all study visits or procedures required by the study protocol, including follow-up visits, and/or fail to comply with all required study procedures;
12. Patients who suffer from any condition or illness that, in the opinion of the Investigator, would compromise patient safety or interfere with the evaluation of the safety of the research drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Complete Molecular Remission | 4 weeks
  Will be estimated along with the 95% credible intervals. Complete molecular response (CMR) was defined as the absence of a detectable BCR-ABL1 transcript with a sensitivity of 0.01%.
Incidence of adverse events (AEs) | 2 years
  Will be graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0. The proportion of patients with AEs will be estimated, along with the Bayesian 95% credible interval.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 2 years
  Will be estimated along with the 95% credible intervals. ORR is defined by Complete Remission (CR)+ CR with incomplete marrow recovery (CRi) .
Duration of Complete Molecular Remission | From the date of acquisition of complete molecular remission until the date of loss of complete molecular remission, assessed up to 2 years.
  Will be estimated along with the 95% credible intervals.
Event-free survival (EFS) | From the first day of treatment until any failure (resistant disease, relapse, or death), assessed up to 2 years
  The Kaplan-Meier method will be used to assess EFS probabilities.
Overall survival (OS) | From the first day of treatment to time of death from any cause, assessed up 2 years
  The Kaplan-Meier method will be used to assess OS probabilities.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Jiangsu Institute of Hematology, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided